CLINICAL TRIAL: NCT03478163
Title: Antibiotics During Intrauterine Balloon Tamponade Placement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems with recruitment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Gregory, Director, Women's Reproductive Health Services, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00051005
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Obstetric Complication; Postpartum Hemorrhage; Postpartum Endometritis
Keywords: Bakri; Intrauterine balloon tamponade; Antibiotics
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Cefazolin; Clindamycin; Injections

STUDY DESIGN:
Intervention Model Description: Open label, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The patient will not receive antibiotics as part of the study, though if at any time her provider chooses to administer antibiotics either prophylactically or for treatment she will not prohibited in any way from this or any other treatment as appropriate.
- Antibiotics (Experimental): The patient will receive a 24-hour course of antibiotics. The primary antibiotic of choice will be cefazolin 1 gm iv q8 hours. If the patient has contraindications to the use of cefazolin including cefazolin allergy, hypersensitivity, or severe beta lactam allergy, then clindamycin 900 mg iv q8 hours will be used instead.
  Interventions: Drug: CeFAZolin 1000 MG; Drug: Clindamycin 900 MG in 6 ML Injection

INTERVENTIONS:
Drug: CeFAZolin 1000 MG — Cefazolin 1000 mg every 8 hours for 3 doses
  Arms: Antibiotics
Drug: Clindamycin 900 MG in 6 ML Injection — Clindamycin 900 mg every 8 hours for 3 doses
  Arms: Antibiotics

SUMMARY:
The goal of this study is to identify whether antibiotics given at the time of placement of an intrauterine balloon tamponade (IBT) will result in reduction of the risk of endometritis. The investigators hypothesize that antibiotics given at the time of intrauterine balloon tamponade will reduce the likelihood of postpartum endometritis.

DETAILED DESCRIPTION:
The investigators will perform a randomized, controlled trial of women who have had a postpartum hemorrhage and received an intrauterine balloon tamponade.

Patients who are candidates for study enrollment will be identified on Labor & Delivery or in the Maternal-Fetal Care Unit. Patients who give consent will be randomized by random number generator to receive either antibiotics (Group A) or no antibiotics (Group B).

If the patient is randomized to Group A, she will receive a 24-hour course of antibiotics. The primary antibiotic of choice will be cefazolin 1 gm iv q8 hours. If the patient has contraindications to the use of cefazolin including cefazolin allergy, hypersensitivity, or severe beta lactam allergy, then clindamycin 900 mg iv q8 hours will be used instead.

If the patient is randomized to Group B, she will not receive antibiotics as part of the study, though if at any time her provider chooses to administer antibiotics either prophylactically or for treatment she will not prohibited in any way from this or any other treatment as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Able to give consent
* Gestational age > 24 weeks
* Postpartum
* Placement of an IBT within the last 2 hours with plans for it to remain in situ for at least 2 hours
* Primary obstetrician amenable to proceeding with either method of management during the study period.

Exclusion Criteria:

* Age < 18 years old
* IBT removed within 2 hours of placement
* Chorioamnionitis
* Insufficient documentation of demographics, delivery outcomes, or peripartum events including postpartum hemorrhage, infectious outcomes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient must be postpartum
Enrollment: 11 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Gregory, MD MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Antibiotics
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Antibiotics | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Full Range); unit: years] | 36 [30 to 41] | 33.83 [27 to 39] | 34.82 [27 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Gravidity [Mean (Full Range); unit: pregnancies] | 3 [2 to 4] | 1.67 [0 to 3] | 2.27 [0 to 4]
Parity [Mean (Full Range); unit: pregnancies] | 1 [0 to 2] | 0.33 [0 to 1] | 0.64 [0 to 2]
Preexisting Hypertension [Count of Participants; unit: Participants] | 0 | 1 | 1
Gestational Hypertension or Preeclampsia [Count of Participants; unit: Participants] | 0 | 0 | 0
Asthma [Count of Participants; unit: Participants] | 0 | 3 | 3
Previous C-section [Count of Participants; unit: Participants] | 4 | 1 | 5
Insurance [Count of Participants; unit: Participants]
  HMO / Managed Care | 2 | 1 | 3
  Military | 0 | 1 | 1
  Private | 3 | 4 | 7
BMI [Mean (Full Range); unit: kg/m^2] — Population: BMI Information for 1/5 control participants unavailable
  kg/m^2
    number analyzed (Participants) | 4 | 6 | 10
    (all) | 35.28 [21.9 to 43.2] | 31.5 [26.2 to 42.5] | 33.01 [21.9 to 43.2]
Multiple Gestation [Count of Participants; unit: Participants] — Population: Multiple gestation information unavailable for 1/5 control participants
  Participants
    number analyzed (Participants) | 4 | 6 | 10
    (all) | 0 | 1 | 1
Gestational Age at Delivery [Mean (Full Range); unit: weeks] — Population: Gestational age information unavailable for 1/5 control participants
  weeks
    number analyzed (Participants) | 4 | 6 | 10
    (all) | 38.25 [37 to 39] | 39.17 [38 to 40] | 38.8 [37 to 40]
Birthweight [Mean (Full Range); unit: grams] — Population: Birthweight information unavailable for 2/5 control participants and 1/6 antibiotics participants
  grams
    number analyzed (Participants) | 3 | 5 | 8
    (all) | 3653.33 [3240 to 3990] | 3632.2 [2965 to 4196] | 3640.13 [2965 to 4196]
Induction [Count of Participants; unit: Participants] — Population: Induction information unavailable for 1/6 antibiotics participants
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 1 | 2 | 3
Labor Augmented by Pitocin [Count of Participants; unit: Participants] — Population: Labor Augmented by Pitocin information unavailable for 1/5 control participants
  Participants
    number analyzed (Participants) | 4 | 6 | 10
    (all) | 2 | 5 | 7
GBS Status [Count of Participants; unit: Participants] — Population: GBS status unavailable for 1/5 control participants
  Participants
    number analyzed (Participants) | 4 | 6 | 10
    Positive GBS Status | 0 | 0 | 0
    Negative GBS Status | 4 | 6 | 10
Mode of Delivery [Count of Participants; unit: Participants]
  Vaginal | 1 | 3 | 4
  Cesarean Section | 4 | 3 | 7
IBT Volume [Mean (Full Range); unit: cc] | 218 [60 to 430] | 273.33 [160 to 360] | 248.18 [60 to 430]
Balloon Deflation: Rapid or Strep [Count of Participants; unit: Participants]
  Rapid | 3 | 6 | 9
  Strep | 2 | 0 | 2
Number of Serial Deflations [Count of Participants; unit: Participants]
  1 Serial Deflations | 3 | 6 | 9
  2 Serial Deflations | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Postpartum Endometritis
Description: Number of participants with postpartum endometritis as defined by clinical documentation
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 3

2. Secondary Outcome: Number of Participants With a Fever
Description: Number of participants with a fever > 38 degrees celsius
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 3

3. Secondary Outcome: Receiving Postpartum Antibiotics
Description: Receiving postpartum antibiotics
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 1 | 3
Participants | 0 | 3

4. Secondary Outcome: Hysterectomy
Description: Hysterectomy
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

5. Secondary Outcome: EBL
Description: Estimated blood loss prior to removal and with IBT in
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: cc
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
cc
  Estimated Blood Loss Pre-IBT | 1626 [1400 to 1800] | 1385.83 [965 to 1800]
  Estimated Blood Loss with IBT in | 165.6 [115 to 295] | 197 [80 to 430]

6. Secondary Outcome: Postpartum Hemoglobin
Description: Postpartum hemoglobin value
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
g/dL | 9.52 [9 to 10.3] | 9.23 [8 to 10.7]

7. Secondary Outcome: Blood Transfusion
Description: Blood transfusions
Time Frame: 2 weeks
Population: Blood transfusion information unavailable for 1/6 antibiotics participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 5
Participants
  0 RBC Transfusions | 3 | 0
  1 RBC Transfusions | 0 | 2
  2 RBC Transfusions | 2 | 2
  3 RBC Transfusions | 0 | 1

8. Secondary Outcome: Maternal ICU Admission
Description: Maternal ICU Admission
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

9. Secondary Outcome: Maternal Death
Description: Maternal death
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

10. Secondary Outcome: Resource Utilization Measures
Description: Duration of admission to maternal-fetal care unit and total hospital admission length of stay
Time Frame: 6 weeks
Population: Duration of admission to maternal-fetal care unit and total hospital admission information unavailable for 1/5 control participants
Measure: Mean (Full Range); unit: hours
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 4 | 6
hours
  MFCU Length of Stay | 29.75 [19 to 53] | 30.67 [20 to 40]
  Total Hospital Length of Stay | 83.75 [71 to 104] | 88.83 [64 to 122]

11. Secondary Outcome: Hospital Readmission
Description: Hospital readmission
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Antibiotics
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Control | Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03478163/Prot_SAP_001.pdf